CLINICAL TRIAL: NCT03329339
Title: 1L Morning-only Polyethylene Glycol Plus Ascorbic Acid With Prepackaged Low-residue Diet Versus 2L Polyethylene Glycol Plus Ascorbic Acid for Bowel Preparation: a Randomized Trial
Brief Title: The Effect of 1L Polyethylene Glycol Plus Ascorbic Acid With Prepackaged Low-Residue Diet for Bowel Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyuk Yoon, Assistant professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-1505-297-003
Record Dates: First submitted 2017-10-09; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Colonoscopy; Colon Polyp; Bowel Preparation Solutions
Keywords: diet
MeSH Terms: conditions — Colonic Polyps | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2 L PEG with ascorbic acid group (No Intervention)
- 1 L PEG with ascorbic acid with PLD (Experimental)
  Interventions: Procedure: 1 L PEG with ascorbic acid with prepackaged, low residue diet

INTERVENTIONS:
Procedure: 1 L PEG with ascorbic acid with prepackaged, low residue diet — Participants who were allocated to the 2 L PEG with ascorbic acid (PEGA) group took 250 ml of PEG with ascorbic acid at 15-min intervals, completing 1 L of the PEG with ascorbic acid protocol at 8:00 PM on the day prior to the procedure. The remaining 1 L of the PEG with ascorbic acid solution was administered in the same manner at 6:00 AM on the day of the procedure. Participants assigned to the 1 L PEG with ascorbic acid with PLD (PLD) group consumed a prepackaged, low residue diet (ZeroCol, Korea Medical Food Inc., Seoul, Korea) which consisted of a breakfast, lunch and dinner, the day prior to colonoscopy. The Participants took 1 L PEG with ascorbic acid solution at 6:00 AM on the day of the colonoscopy in the same way as described above. All of the subjects ingested 500 mL of water for every 1 L of 1 L PEG with ascorbic acid solution consumed. The Participants completed all of the administrations at least 2 hours before the colonoscopy.
  Arms: 1 L PEG with ascorbic acid with PLD

SUMMARY:
Background 2L polyethylene glycol plus ascorbic acid (PEGA) is known to be as effective as standard 4L polyethylene glycol for bowel preparation. However, the volume of this regimen is still large. Therefore, the present investigators evaluated the potential of 1L PEGA with prepackaged low-residue diet (PLD) for an alternative to 2L PEGA.

Aim: To evaluate efficacy of 1L PEG with ascorbic acid combined with prepackaged low-residue diet as bowel preparation for colonoscopy.

Methods: The subjects were randomly assigned to either groups. PEGA group received 2L PEGA split regimen. PLD group received PLD on the day preceding colonoscopy and 1L PEGA on the morning of colonoscopy. One blinded physician performed colonoscopy and evaluated the degree of bowel preparation using Boston bowel preparation score (BBPS). A questionnaire regarding tolerability and safety were also gathered.

ELIGIBILITY:
Inclusion Criteria:

* anyone who were scheduled for an outpatient colonoscopy below indication

  1. patient who need colonic polyp screening
  2. patient who have hematochezia
  3. patient who have fecal occult blood test positive result

Exclusion Criteria:

* ileus
* inflammatory bowel disease-
* gastrointestinal malignancy
* severe cardiac disease (heart failure beyond NYHA Class III)
* chronic obstructive pulmonary disease,
* decompensated liver cirrhosis; coagulopathy
* Female patients with pregnant or breastfeeding.
* who use long-term use of sedative, anti-spasmodic, prokinetic, laxative or anti-diarrheal medications

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Achievement of preparation adequacy | assessed at the colonoscopy day
  Definition: Achievement of preparation adequacy was defined by as having BBPS scores of 2 or 3 for all colon segments.
  BBPS was measured by Physician who performing colonoscopy. To maintain precise evaluation, the physician participated in an online training program from www.cori.org/bbps. For each colon segment, BBPS preparation score ranged 0 to 3. Definition of BBPS are presented at www.cori.org/bbps

SECONDARY OUTCOMES:
Tolerability and adverse events | assessed at the colonoscopy day
  Tolerability and adverse events were measured by comprehensive questionnaire. Participants were asked about the presence of distressing symptoms, such as abdominal pain/discomfort or nausea/vomiting, and if they had problems taking the entire dose. The subjects also reported the percentage of the preparation they completed (100%, 90~99%, <90%), regardless of solution or meals. Adverse events are categorized by CTCAE v4.03.

REFERENCES:
- [Derived] Lee JW, Choi JY, Yoon H, Shin CM, Park YS, Kim N, Lee DH. Favorable outcomes of prepackaged low-residue diet on bowel preparation for colonoscopy: Endoscopist-blinded randomized controlled trial. J Gastroenterol Hepatol. 2019 May;34(5):864-869. doi: 10.1111/jgh.14499. Epub 2018 Oct 24. PMID 30278110